CLINICAL TRIAL: NCT03212430
Title: The Effect of Intravenous L-kynurenine (LKYN) on Cerebral Hemodynamics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: L-kynurenin H-16033148
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Headache
Keywords: L-kynurenine; Cerebral hemodynamic; Headache; Mohammad Al-Mahdi Al-Karagholi
MeSH Terms: conditions — Headache | interventions — Kynurenine

STUDY DESIGN:
Intervention Model Description: Pilot, Open label
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: L-kynurenine — intravenous infusion of L-kynurenine to healthy individuals.

SUMMARY:
To measure the cerebral hemodynamic effect of L-kynurenine.

DETAILED DESCRIPTION:
Aim: To investigate the physiological effect of L-Kynurenine after intravenous administration to healthy volunteers.

Hypothesis: L-kynurenine induces vasodilation in the cerebral vessels and trigger headache in healthy individuals.

Methods: 6 healthy volunteers will receive intravenous infusion of L-kynurenine using the following doses 50 microgram/kg, 100 microgram/kg, 150 microgram/kg, 300 microgram/kg, 500 microgram/kg, 1 mg/kg and 5 mg/kg over 20 min on 7 different days with at least 1 day in between. Before and after infusion (at 20, 40, 60, 80 and 100 min) we will record vital signs, circumferences of middle cerebral artery, superficial temporalis artery and headache intensity and characteristics.

The subjects will then have a questionnaire about headache for the following 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes.
2. 18-60 years.
3. 50-90 kg.
4. Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

1. All primary headaches
2. First-degree relative with migraine
3. Headache less than 48 hours before the tests start
4. Daily consumption of drugs of any kind other than oral contraceptives.
5. Pregnant or nursing women. Cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Velocity of MCA (VMCA) | Change from baseline VMCA at two hours after administration of L-kynurenine
  Measured in MCA (middle cerebral artery) bilaterally with ultrasound (TCD) (2 Mhz, DWL)
The diameter of the STA (superficial temporal artery) | Change from baseline VMCA at two hours after administration of L-kynurenine
  Measured by high-frequency ultrasound 12 of 29 (Derma Scan C, Cortex Technology, Denmark)
Headache | occurrence of headache undtil 24 hours after infusion.
  Headache declared orally on a verbal rating scale (VRS) 0-10. 0 represents no pain and 10 the worst possible headache.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Professor, Principal Investigator — Professor of neurology
Locations (1):
- Rigshospitalet-Glostrup, Glostrup Municipality, Nordre Ringvej 57, Denmark

IPD SHARING:
Plan to Share IPD: Yes
1. Using a controlled access approach, using a transparent and robust system to review requests and provide secure data access; 2. seeking consent for sharing IPD from trial participants in all future clinical trials with adequate assurance that patient privacy and confidentiality can be maintained; and 3. Establishing an approach to resource the sharing of IPD which would include support from trial funders, sponsor organisations and users of IPD